CLINICAL TRIAL: NCT06620861
Title: Investigation on a New Power Knee Firmware Update on Gait and Daily Life Activities, a Randomized Controlled Double-blinded Cross-over Investigation
Brief Title: Investigation on a New Power Knee Firmware Update on Gait and Daily Life Activities for Transfemoral Amputees
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more data collection needed under this protocol
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CIP2024070123
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Amputation; Transfemoral Amputation
Keywords: Microprocessor knee; prosthesis; powered prosthesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Other): Group A will start with the current marketed firmware.
  Interventions: Device: Power Knee Firmware Update; Device: Power Knee Current Marketed Firmware
- Group B (Other): Group B will start with the firmware in development.
  Interventions: Device: Power Knee Firmware Update; Device: Power Knee Current Marketed Firmware

INTERVENTIONS:
Device: Power Knee Firmware Update — The firmware in development will be uploaded to the device.
Device: Power Knee Current Marketed Firmware — The current marketed firmware will be uploaded to the device.

SUMMARY:
The goal of this interventional study is to investigate a new firmware in development for Power Knee on gait and daily life activities in unilateral transfemoral amputees. The main question it aims to answer is:

What are the effects of a new firmware on sit-to-stand, level walking and stair ascent ?

Researchers will compare both a new and the current marketed firmware to see if there is any changes in performance.

Participants will be asked to perform some activities of daily living and some functional tests.

ELIGIBILITY:
Inclusion Criteria:

* 50 kg < body weight < 116 kg
* lower limb loss, amputation or deficiency
* cognitive ability to understand all instructions and questionnaires in the study
* Unilateral transfemoral amputees that are regular Power Knee users for at least 4 weeks
* age ≥ 18 years
* Moderate to high active subjects
* Willing and able to participate in the study and follow the protocol
* Comfortable and stable socket fit
* No socket issues/changes in the last 6 weeks

Exclusion Criteria:

* Users with pain
* Bilateral amputees
* Users using passive microprocessor controlled knees
* Users with cognitive impairment
* Users with co-morbidities in the contra lateral limb, which affect their functional mobility
* Hip disarticulation amputees
* Users with osseointegrated prosthesis
* Pregnant users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete Simpson, Principal Investigator — Össur Americas
Locations (1):
- Oakland Orthopedic Appliances Inc, Bay City, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This is proprietary data as part as the investigation.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects with transfemoral amputation provided informed consent and were formally enrolled in the study, as reflected in the Protocol Section (6). However, one enrolled subject did not proceed to randomization due to low activity level and fatigue, and therefore did not start the intervention. As a result, only 5 participants were assigned to an Arm/Group and included in the Participant Flow module (5), and their data are presented in the Baseline Characteristics and analysis.
Groups:
- Current Marketed Firmware Before New Firmware: Group A will start with the current marketed firmware.
  Power Knee Firmware Update: The firmware in development will be uploaded to the device.
  Power Knee Current Marketed Firmware: The current marketed firmware will be uploaded to the device.
- New Firmware Before Current Marketed Firmware: Group B will start with the firmware in development.
  Power Knee Firmware Update: The firmware in development will be uploaded to the device.
  Power Knee Current Marketed Firmware: The current marketed firmware will be uploaded to the device.
Period: Overall Study
Arm/Group | Current Marketed Firmware Before New Firmware | New Firmware Before Current Marketed Firmware
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject did not complete the protocol and were not randomized in a group due to a low activity level and some fatigue. Hence, their data is not analyzed, only five subjects were included in the data analysis.
Groups:
- Combined Crossover Evaluation Group: For the analysis, data from both participant groups were pooled. Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware.
  Power Knee Firmware Update: The investigational (new) firmware was installed on the device.
  Power Knee Current Marketed Firmware: The existing marketed firmware was installed on the device.
  In Group A, participants first used the current marketed firmware before switching to the investigational firmware.
  In Group B, participants first used the investigational firmware before switching to the current marketed firmware.
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject did not complete the protocol and were not randomized in a group due to a low activity level and some fatigue. Hence, their data is not analyzed, only five subjects were included in the data analysis.
  years | 55.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject did not complete the protocol and were not randomized in a group due to a low activity level and some fatigue. Hence, their data is not analyzed, only five subjects were included in the data analysis.
  Participants
    Female | 2
    Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Amputation level Transfemoral [Count of Participants; unit: Participants] — Population: One subject did not complete the protocol and were not randomized in a group due to a low activity level and some fatigue. Hence, their data is not analyzed, only five subjects were included in the data analysis.
  Participants | 5

OUTCOME MEASURES:

1. Primary Outcome: Sit to Stand Activity
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing sit to stand activity
Time Frame: after acclimatization at day 1 during the single study event
Measure: Count of Participants; unit: Participants
Groups:
- Combined Crossover Evaluation Group: For the analysis, data from both participant groups were pooled. Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware.
  Power Knee Firmware Update: The investigational (new) firmware was installed on the device.
  Power Knee Current Marketed Firmware: The existing marketed firmware was installed on the device.
  In Group A, participants first used the current marketed firmware before switching to the investigational firmware.
  In Group B, participants first used the investigational firmware before switching to the current marketed firmware.In Group B, participants initially used the investigational firmware, and then switched to the current marketed firmware.
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 5
Participants
  worse | 1
  similar | 1
  better | 3

2. Primary Outcome: Stand to Sit Activity
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing stand to sit activity
Time Frame: after acclimatization at day 1 during the single study event
Measure: Count of Participants; unit: Participants
Groups:
- Combined Crossover Evaluation Group: For the analysis, data from both participant groups were pooled. Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware.
  Power Knee Firmware Update: The investigational (new) firmware was installed on the device.
  Power Knee Current Marketed Firmware: The existing marketed firmware was installed on the device.
  In Group A, participants first used the current marketed firmware before switching to the investigational firmware.
  In Group B, participants first used the investigational firmware before switching to the current marketed firmware.
  In Group B, participants initially used the investigational firmware, and then switched to the current marketed firmware.
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 5
Participants
  worse | 1
  similar | 3
  better | 1

3. Primary Outcome: Level Ground Walking
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing level ground walking.
Time Frame: after acclimatization at day 1 during the single study event
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 5
Participants
  worse | 2
  similar | 1
  bettter | 2

4. Other Pre Specified Outcome: 2MWT
Description: The 2-Minute Walk Test is a clinical assessment used to measure an individual's walking endurance and functional capacity. During the test, the participant is instructed to walk for 2 minutes at their comfortable pace along a marked course. The total distance walked within the 2-minute period is recorded (in meters).
Time Frame: after acclimatization at day 1 during the single study event
Population: Only 2 subjects performed this test.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Current Marketed Firmware: Results obtained with the current marketed firmware.
- New Investigational Firmware: Results obtained with the new investigational firmware.
Arm/Group | Current Marketed Firmware | New Investigational Firmware
Number analyzed (Participants) | 2 | 2
meters | 173.5 (19.1) | 179.5 (0.7)

5. Other Pre Specified Outcome: 10mWT
Description: The 10-Meter Walk Test is a commonly used clinical assessment to measure an individual's walking speed over a short distance. During the test, the participant is asked to walk a distance of 10 meters at their fastest possible pace. The time taken to walk the 10 meters is recorded.
Time Frame: after acclimatization at day 1 during the single study event
Population: Only 4 subjects performed this test.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Current Marketed Firmware | New Investigational Firmware
Number analyzed (Participants) | 4 | 4
seconds | 6.91 (1.14) | 6.61 (1.66)

6. Other Pre Specified Outcome: Stair Ascent Activity
Description: Stair assessment index (0-13)
Time Frame: after acclimatization at day 1 during the single study event
Population: Data for stair ascent activities (Outcome Measures 6-9) could not be reported because these activities were not tested during the study. The investigational firmware was not finalized in time for stair ascent, and therefore this activity was not included in the testing protocol. As a result, no data were collected for these Outcome Measures. In the protocol, data related to stair ascent was considered exploratory.
Groups:
- Combined Crossover Evaluation Group: For the analysis, data from both arms were combined.
  Power Knee Firmware Update: The firmware in development will be uploaded to the device.
  Power Knee Current Marketed Firmware: The current marketed firmware will be uploaded to the device.
  In Group A, participants initially used the current marketed firmware, and then switched to the investigational firmware.
  In Group B, participants initially used the investigational firmware, and then switched to the current marketed firmware.
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Entering Stair Ascent Mode
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing stair ascent (entering) activity
Time Frame: after acclimatization at day 1 during the single study event
Population: as for outcome 6
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Exiting From Stair Ascent Mode
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing the stair ascent (exiting) activity.
Time Frame: after acclimatization at day 1 during the single study event
Population: as for outcome 6
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Perception of Stair Ascent Activity
Description: Each participant rated whether the new investigational firmware was worse, similar, or better compared to the current marketed firmware when performing stair ascent activity
Time Frame: after acclimatization at day 1 during the single study event
Population: as for outcome 6
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Current Marketed Firmware Before New Firmware | New Firmware Before Current Marketed Firmware
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT06620861/Prot_SAP_001.pdf